CLINICAL TRIAL: NCT01202253
Title: A Study To Describe The Early Clinical Experience With Anidulafungin In Patients With Liver Disease At King's College Hospital NHS Trust, London
Brief Title: Early Clinical Experience With Anidulafungin In Patients With Liver Disease In The United Kingdom
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A8851028
Record Dates: First submitted 2010-09-13; First posted 2010-09-15 (Estimated); Results first posted 2012-10-11 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Candidiasis
Keywords: Ecalta; Eraxis; Candida; Candidemia; Systemic Candidiasis; ICU; Intensive Care Unit; Critical Care Unit
MeSH Terms: conditions — Candidiasis; Torulopsis; Candidemia; Systemic candidiasis | interventions — Anidulafungin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Anidulafungin
  Interventions: Drug: anidulafungin

INTERVENTIONS:
Drug: anidulafungin — A single 200 mg loading dose should be administered on Day 1, followed by 100 mg daily thereafter.
  Other Names: ECALTA, ERAXIS

SUMMARY:
The purpose of this study is to describe the real world effectiveness of anidulafungin in clinical practice in a large Liver Unit in the United Kingdom.

DETAILED DESCRIPTION:
All subjects that have been treated with Anidulafungin according to its licence during the period of July 2009 and September 2010 will be included.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been prescribed anidulafungin between 1st July 2009 and 30th September 2010.

Patients admitted to specialist liver unit wards and the Liver Intensive Therapy Unit during this period

Exclusion Criteria:

* Patients who participated in any interventional clinical trial during this episode of sepsis.

Patients who received anidulafungin for infection prophylaxis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects admitted with candidiasis infections to the Liver Unit at King's College Hospital (United Kingdom) who are prescribed anidulafungin.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, London, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8851028&StudyName=Early%20Clinical%20Experience%20With%20Anidulafungin%20In%20Patients%20With%20Liver%20Disease%20In%20The%20United%20Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Anidulafungin: Anidulafungin (Ecalta) 200 milligram (mg) intravenous infusion on the first day followed by 100 mg intravenous infusion once daily as per investigator's discretion.
Period: Overall Study
Arm/Group | Anidulafungin
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
Age, Customized [Mean (Inter-Quartile Range); unit: years] | 50.5 (16.4) [36.4 to 63.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Percentage of participants with elective or emergency hospital admission [Number; unit: percentage of participants]
  Elective admission | 72
  Emergency admission | 28
Overall duration of hospital stay [Mean (Inter-Quartile Range); unit: days] | 86.46 [50.00 to 99.50]
Number of participants with underlying liver disease [Number; unit: participants]
  Acute liver disease | 1
  Chronic liver disease | 8
  Chronic and acute liver disease | 3
  Hepatopancreaticobiliary disease | 12
  Hepatopancreaticobiliary disease, pancreatitis | 3
  Liver transplant | 4
  Liver transplant, acute liver disease | 3
  Liver transplant, acute liver failure | 1
  Liver transplant, acute liver disease, failure | 1
  Liver transplant, chronic liver disease | 11
  Liver transplant, chronic disease, acute failure | 1
  Liver transplant, chronic disease, pancreatitis | 1
  Liver laceration | 1
Number of participants with relevant co-morbidities [Number; unit: participants] — Other co-morbidities included renal failure or impairment, multi-organ failure, previous liver transplants, liver abscess and hepatic artery thrombosis.
  participants
    History of alcohol abuse | 19
    Diabetes | 18
    Hepatitis C | 5
    Malignancy | 12
    Other | 37
Number of participants with markers of illness severity [Number; unit: participants]
  Upper gastrointestinal (GI) bleed | 21
  Central line of admission | 25
  Total parenteral nutrition | 26
  Intubated on admission | 15
  Major surgery | 37
  Renal failure | 31
Percentage of participants with Model for End-Stage Liver Disease (MELD) score [Number; unit: percentage of participants] — MELD is a scoring system for assessing the severity of chronic liver disease. MELD uses the participant's values for serum bilirubin, serum creatinine, and the INR for prothrombin time to predict survival. In interpreting the MELD score in hospitalized participants, the 3 month mortality is: greater than or equal to 40 - 71.3% mortality; 30-39 - 52.6% mortality; 20-29 - 19.6% mortality; 10-19 - 6.0% mortality; less than 10 - 1.9% mortality.
  percentage of participants
    Less than 10 | 7
    10 to 19 | 13
    20 to 29 | 37
    30 to 39 | 37
    Greater than or equal to 40 | 7
Number of participants with disease severity score [Number; unit: participants] — Disease severity score was based on acute physiological assessment and chronic health evaluation (APACHE), used for assessing severity of illness in acutely ill participants in intensive care units (ICUs). Total possible score range: 0 to 71 where higher score represented higher predicted mortality.
  participants | NA — Data was not analyzed as the study was retrospective and disease severity score was not available for the participants.
Number of participants with total white cell count [Number; unit: participants]
  Less than 4 * 10^9/Liter | 8
  4 to 11 * 10^9/Liter | 3
  Greater than 11 * 10^9/Liter | 39
Number of participants with International Normalized Ratio (INR) results [Number; unit: participants] — Prothrombin time is a measure of the extrinsic pathway of coagulation that is used to determine the clotting tendency of blood. INR is the ratio of a participant's prothrombin time to a normal (control) sample.
  participants
    Less than 0.8 | 0
    0.8 to 1.6 | 32
    Greater than 1.6 | 18
Number of participants with C-reactive protein (CRP) levels [Number; unit: participants] — CRP levels were categorized either less than 5 mg/L and greater than or equal to 5 mg/L. Those participants with CRP levels not analyzed were reported under 'not done' category.
  participants
    Less than 5 mg/liter (mg/L) | 2
    Greater than or equal to 5 mg/L | 44
    Not done | 4
Number of participants with urea levels [Number; unit: participants]
  Less than 3.3 millimole/Liter (mmol/L) | 1
  3.3 to 6.7 mmol/L | 15
  Greater than 6.7 mmol/L | 34
Percentage of participants with creatinine clearance outside normal range [Number; unit: percentage of participants] — Normal values for creatinine clearance for an adult are below 80 milliliter/minute (mL/min).
  percentage of participants | NA — Data was not analyzed as the study was retrospective and data for creatinine clearance was not available for the participants.
Percentage of participants prescribed with immunosuppressant drugs [Number; unit: percentage of participants]
  Azathioprine | 2
  Ciclosporin | 2
  Methylprednisolone | 2
  Prednisolone | 44
  Tacrolimus or tacrolimus modified release (MR) | 50
Percentage of participants prescribed with concomitant systemic antifungals [Number; unit: percentage of participants]
  Amphotericin | 2
  Fluconazole | 12
Percentage of participants prescribed with concomitant antibiotics [Number; unit: percentage of participants]
  Amikacin | 22
  Ciprofloxacin | 2
  Clarithromycin | 2
  Colistin | 4
  Co-trimoxazole | 8
  Erythromycin | 4
  Gentamicin | 4
  Linezolid | 28
  Metronidazole | 4
  Tazocin | 34
  Vancomycin | 38
Number of participants with concomitant antibiotics prescribed [Number; unit: participants] — Participants were categorized into 6 categories, 0 to 5 based on the number of concomitant antibiotics prescribed to them.
  participants
    0 antibiotic | 4
    1 antibiotic | 8
    2 antibiotics | 22
    3 antibiotics | 8
    4 antibiotics | 7
    5 antibiotics | 1
Duration of antibiotic course [Median (Inter-Quartile Range); unit: days] | 16.00 [11.00 to 21.75]
Percentage of participants prescribed with antiviral courses [Number; unit: percentage of participants]
  Aciclovir | 2
  Ganciclovir | 6
  Oseltamivir | 2
  Valganciclovir | 20
Duration of antiviral courses [Median (Inter-Quartile Range); unit: days] | NA [NA to NA] — Data was not analyzed as the study was retrospective and duration of antiviral courses was not available for the participants.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Favorable Outcome
Description: Favorable outcome was defined as favorable clinical response and documented or presumed microbial eradication (two negative follow-up blood cultures for bloodstream infections or a successful clinical response without follow-up cultures for other infections). Favorable clinical response was defined as clinical resolution of signs and symptoms of infection and no need to change or add to antifungal therapy, or transition to oral antifungal to complete therapy.
Time Frame: Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria. Here, 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 46
percentage of participants | 76.1 [64.3 to 87.9]

2. Secondary Outcome: Percentage of Participants With Unfavorable Outcome
Description: Unfavorable outcome was defined as the need to change to another antifungal agent because of lack of clinical response or death due to the antifungal infection or microbiologic persistence of the fungus or superinfection with a new Candida, Aspergillus or other fungal strain occurring at least 3 days and up to 14 days of anidulafungin therapy, or a lack of follow up data about clinical and microbiologic responses at the end of anidulafungin therapy.
Time Frame: Day 28 post-treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 46
percentage of participants | 23.9 [12.1 to 35.7]

3. Secondary Outcome: Percentage of Participants Who Died Due to All Causes
Description: Death due to all causes included death attributable to fungal infection, death unrelated to fungal infection and death due to multiple causes.
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 38.0 [24.5 to 51.5]

4. Secondary Outcome: Percentage of Participants With Death Attributable to Fungal Infection
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 0 [0 to 0]

5. Secondary Outcome: Percentage of Participants With Death Unrelated to Fungal Infection
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 36.0 [22.7 to 49.3]

6. Secondary Outcome: Percentage of Participants With Favorable Clinical Response
Description: Favorable clinical response was defined as clinical resolution of signs and symptoms of infection and no need to change or add to antifungal therapy, or transition to oral antifungal to complete therapy.
Time Frame: Day 28 post-treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 46
percentage of participants | 80.4 [69.4 to 91.4]

7. Secondary Outcome: Percentage of Participants With Lack of Clinical Response
Description: as for outcome 6
Time Frame: Day 28 post-treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 46
percentage of participants | 19.6 [8.6 to 30.6]

8. Secondary Outcome: Percentage of Participants Requiring Change or Additional Antifungal Therapy
Description: Lower limit of confidence interval was reported as 0 if the same was calculated as less than 0 by standard calculations (outside the valid range of 0 to 100).
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants
  Due to all reasons | 16.0 [5.8 to 26.2]
  Due to lack of clinical response | 4.0 [0.0 to 9.4]
  Due to adverse event | 0.0 [0.0 to 0.0]

9. Secondary Outcome: Percentage of Participants With Oral Antifungal Started to Complete Therapy
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 32.0 [19.1 to 44.9]

10. Secondary Outcome: Percentage of Participants With Documented Eradication of Infecting Species
Description: Documented microbial eradication was defined as 2 negative follow-up blood cultures for bloodstream infections.
Time Frame: Baseline
Population: Data was not analyzed as the study was retrospective and data for eradication of candida infection was not documented in the participants' medical notes.
Arm/Group | Anidulafungin
Number analyzed (Participants) | 0

11. Secondary Outcome: Percentage of Participants With Resolution of Signs of Infection According to Ultrasound Scan Results
Description: An ultrasound scan was performed and the resultant scan was reviewed for the presence of the infection as per investigator's discretion.
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 80.0 [68.9 to 91.1]

12. Secondary Outcome: Percentage of Participants With Resolution of Signs of Infection According to Computerized Tomography (CT) Scan Results
Description: A CT scan was performed and the resultant scan was reviewed for the presence of the infection as per investigator's discretion.
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 68.0 [55.1 to 80.9]

13. Secondary Outcome: Percentage of Participants With Abnormal Results for Liver Function at Initiation of Drug Therapy
Description: Percentage of participants with abnormal liver function results were based on 4 liver function variables- bilirubin, aspartate transaminase, alkaline phosphatase and gamma glutamyl transferase. Normal reference ranges of these variables are: plasma bilirubin: 3-17 micromoles/L or 2.5-10 mg/L for adults; aspartate transaminase: 6-34 International Units/Liter (IU/L) for females and 8-40 IU/L for males; alkaline phosphatase: 5-38 IU/L for females and 10-50 IU/L for males; gamma glutamyl transferase: 7-32 IU/L for females and 11-50 IU/L for males. Upper limit of confidence interval was reported as 100 if the same was calculated as greater than 100 by standard calculations (outside the valid range of 0 to 100).
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 98.0 [94.1 to 100.0]

14. Secondary Outcome: Percentage of Participants With Abnormal Results for Liver Function at End of Drug Therapy
Description: Percentage of participants with abnormal liver function results were based on 4 liver function variables- bilirubin, aspartate transaminase, alkaline phosphatase and gamma glutamyl transferase. Normal reference ranges of these variables are: plasma bilirubin: 3-17 micromoles/L or 2.5-10 mg/L for adults; aspartate transaminase: 6-34 IU/L for females and 8-40 IU/L for males; alkaline phosphatase: 5-38 IU/L for females and 10-50 IU/L for males; gamma glutamyl transferase: 7-32 IU/L for females and 11-50 IU/L for males.
Time Frame: Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 74.0 [61.8 to 86.3]

15. Secondary Outcome: Percentage of Participants With Liver Function Test Results at Least Twice the Baseline Value During Period of Drug Therapy
Description: Percentage of participants with liver function test results at least twice the baseline value during period of drug therapy was calculated for the liver function variables, bilirubin, aspartate transaminase, alkaline phosphatase and gamma glutamyl transferase.
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants
  Bilirubin test | 24.0 [12.2 to 35.8]
  Aspartate transaminase test | 40.0 [26.4 to 53.6]
  Alkaline phosphatase test | 34.0 [20.9 to 47.1]
  Gamma glutamyl transferase test | 36.0 [22.7 to 49.3]

16. Secondary Outcome: Percentage of Participants With Creatinine Clearance at Least Twice the Baseline Value During Period of Drug Therapy
Time Frame: Baseline up to Day 28 post-treatment
Population: Data was not analyzed as the study was retrospective and data for creatinine clearance was not available for the participants.
Arm/Group | Anidulafungin
Number analyzed (Participants) | 0

17. Secondary Outcome: Percentage of Participants Admitted to Liver Intensive Therapy Unit (LITU)
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 78.0 [66.5 to 89.5]

18. Secondary Outcome: Duration of Stay at Liver Intensive Therapy Unit (LITU)
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure.
Measure: Mean (Inter-Quartile Range); unit: days
Arm/Group | Anidulafungin
Number analyzed (Participants) | 39
days | 29.38 [7.00 to 38.00]

19. Secondary Outcome: Percentage of Participants With Absolute Neutrophil Count Less Than 500 Per Cubic Millimeter (/mm^3) and Greater Than or Equal to 500 /mm^3
Description: Lower limit of confidence interval was reported as 0 if the same was calculated as less than 0 and upper limit of confidence interval was reported as 100 if the same was calculated as greater than 100, by standard calculations (outside the valid range of 0 to 100).
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants
  Less than 500/mm^3 | 2.0 [0.0 to 5.9]
  Greater than or equal to 500/mm^3 | 98.0 [94.1 to 100.0]

20. Secondary Outcome: Percentage of Participants With Concomitant Bacterial or Viral Infection
Description: Upper limit of confidence interval was reported as 100 if the same was calculated as greater than 100 by standard calculations (outside the valid range of 0 to 100).
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants
  Bacterial infection | 96.0 [90.6 to 100.0]
  Viral infection | 46.0 [32.2 to 59.8]

21. Secondary Outcome: Percentage of Participants Prescribed With Systemic Antifungal Within 30 Days Before Study Start
Description: as for outcome 8
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants
  Amphotericin | 4.0 [0.0 to 9.4]
  Caspofungin | 4.0 [0.0 to 9.4]
  Fluconazole | 70.0 [57.3 to 82.7]

22. Secondary Outcome: Dose Changes for Immunosuppressant Drugs
Time Frame: Baseline up to Day 28 post-treatment
Population: Data was not analyzed as the study was retrospective and data for dose change for immunosuppressant drugs was not available.
Arm/Group | Anidulafungin
Number analyzed (Participants) | 0

23. Secondary Outcome: Percentage of Participants With Probable or Proven Fungal Infection at the Initiation of Drug Therapy
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants
  Probable fungal infection | 28.0 [15.6 to 40.4]
  Proven fungal infection | 72.0 [59.6 to 84.4]

24. Secondary Outcome: Percentage of Participants With Documented Body Temperature Above 38.0 Degree Celsius or Below 36.0 Degree Celsius Within 24 Hour Period Prior to Initiation of Drug Therapy
Description: as for outcome 19
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants
  Above 38.0 degree Celsius | 98.0 [94.1 to 100.0]
  Below 36.0 degree Celsius | 2.0 [0.0 to 5.9]

25. Secondary Outcome: Percentage of Participants With Systolic Blood Pressure More Than 2 Standard Deviations Below the Mean for Age Recorded Within 24 Hour Period Prior to Initiation of Drug Therapy
Description: as for outcome 8
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 4.0 [0.0 to 9.4]

26. Secondary Outcome: Number of Participants With Infection Sites as Per Microbiological Analysis
Description: Infection sites included blood, chest, urinary tract, intra-abdominal, bile duct, liver, kidney, mouth and esophagus.
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
participants
  Blood only | 4
  Blood and chest | 1
  Blood and urinary tract | 2
  Chest only | 3
  Intra-abdominal | 13
  Intra-abdominal and bile duct | 3
  Intra-abdominal and blood | 4
  Intra-abdominal, chest and liver | 1
  Intra-abdominal and kidney | 1
  Intra-abdominal and liver | 2
  Liver only | 1
  Liver and urinary tract | 1
  Esophagus and mouth | 1
  Urinary tract and chest | 1
  Urinary tract and esophagus | 1

27. Secondary Outcome: Number of Participants With Infection Sites as Per Ultrasound Scan and Computerized Tomography (CT) Scan
Time Frame: Baseline
Population: Data was not analyzed as the study was retrospective and data for infection site as per ultrasound and CT scan was not available.
Arm/Group | Anidulafungin
Number analyzed (Participants) | 0

28. Secondary Outcome: Infecting Organisms by Species
Time Frame: Baseline up to Day 14 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
participants
  Candida albicans | 17
  Candida glabrata | 17
  Candida guilliermondii | 3
  Candida krusei | 2
  Candida parapsilosis | 3
  Candida species (spp) | 16
  Candida spp (non Candida albicans) | 1
  Candida tropicalis | 1
  Fusarium dimerum | 1
  Saccharomyces cerevisiae | 2
  Yeast | 2
  Adenovirus | 1
  Citrobacter | 2
  Clostridium difficile | 3
  Cytomegalovirus (CMV) | 9
  Escherichia coli | 5
  Escherichia faecalis | 4
  Escherichia faecium | 4
  Epstein-Barr virus (EBV) | 3
  Elizabeth meningoseptica cum chrysobacterium | 1
  Enterobacter cloacae | 1
  Enterobacter spp | 3
  Hemagglutinin 1 Neuraminidase 1 (H1N1)- swine flu | 3
  Herpes simplex virus type 1 | 2
  Klebsiella oxytoca | 1
  Klebsiella pneumonia | 1
  Klebsiella spp | 4
  Methicillin-resistent Staphylococcus aureus | 1
  Pneumocystic jiroveci | 1
  Pseudomonas spp | 5
  Respiratory syncytial virus | 1
  Rhinovirus | 1
  Staphylococcus aureus | 3
  Staphylococcus capitis | 1
  Stenotrophomonas maltophilia | 1
  Stenotrophomonas spp | 3
  Vancomycin-resistant enterococcus | 7
  Pseudomonas aeruginosa | 1
  Staphylococcus epidermidis | 1

29. Secondary Outcome: Percentage of Participants With Prior Colonization With Candida by Species
Description: as for outcome 8
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants
  Candida albicans | 16.0 [5.8 to 26.2]
  Candida glabrata | 10.0 [1.7 to 18.3]
  Candida guilliermondii | 2.0 [0.0 to 5.9]
  Candida spp | 12.0 [3.0 to 21.0]
  Candida tropicalis | 2.0 [0.0 to 5.9]
  Candida species unknown | 6.0 [0.0 to 12.6]

30. Secondary Outcome: Percentage of Participants With Prior Colonization With Candida by Colonization Index
Time Frame: Baseline
Population: Data for prior colonization by colonization index was not analyzed as the study was retrospective and colonization index was not recorded for the participants.
Arm/Group | Anidulafungin
Number analyzed (Participants) | 0

31. Secondary Outcome: Percentage of Participants With Other Prior Fungal Infection by Species and Colonization Index
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 0

32. Secondary Outcome: Number of Participants Who Received Water-based and Ethanol-based Formulation
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
participants
  Water based formulation | 16
  Ethanol based formulation | 34

33. Secondary Outcome: Percentage of Participants Who Received Water-based and Ethanol-based Formulation
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants
  Water based formulation | 32.0 [19.1 to 44.9]
  Ethanol based formulation | 68.0 [55.1 to 80.9]

34. Secondary Outcome: Percentage of Participants Who Received 200 mg Loading Dose
Time Frame: Day 1
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 100.0 [100.0 to 100.0]

35. Secondary Outcome: Percentage of Participants Who Received 100 mg Dose on Day 2
Time Frame: Day 2
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 100.0 [100.0 to 100.0]

36. Secondary Outcome: Percentage of Participants Who Received 200 mg Dose on Day 1 and 100 mg for All Subsequent Doses
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 100.0 [100.0 to 100.0]

37. Secondary Outcome: Number of Participants With Other Dosing Patterns
Description: The other dosing patterns for anidulafungin included any dosing pattern different from 200 mg loading dose on Day 1 followed by 100 mg doses subsequently starting from Day 2.
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
participants | 0

38. Secondary Outcome: Duration of Anidulafungin Therapy
Time Frame: Baseline
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
days | 17.96 (11.04)

39. Secondary Outcome: Number of Serious Adverse Events (SAEs)
Description: Any untoward medical occurrence in a participant who received study treatment was considered an adverse event (AE) without regard to possibility of causal relationship. An AE resulting in any of the following outcomes, or deemed to be significant for any other reason, was considered to be a SAE: death; initial or prolonged inpatient hospitalization; a life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number; unit: events
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
events | 5

40. Secondary Outcome: Percentage of Participants With One or More Drug-related Serious Adverse Events (SAEs)
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number; unit: percentage of participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
percentage of participants | 0

41. Secondary Outcome: Number of Participants With Different Types of Drug-related Serious Adverse Events
Time Frame: Baseline up to Day 28 post-treatment
Population: Full analysis set included all participants who met the defined eligibility criteria.
Measure: Number; unit: participants
Arm/Group | Anidulafungin
Number analyzed (Participants) | 50
participants | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Anidulafungin
Serious Adverse Events (participants affected / at risk) | 5/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anidulafungin (N=50)
New Candida parapsilosis infection (General disorders) | 1
Breakthrough Candida glabrata infection (General disorders) | 2
Breakthrough Candida parapsilosis infection (General disorders) | 1
Continuing Candida glabrata infection (General disorders) | 1

LIMITATIONS AND CAVEATS:
Protocol-specified endpoint, percentage of participants with presumed eradication of infecting species, was not presented as a separate outcome measure because the 'presumed eradication' was considered same as favorable clinical response.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.